CLINICAL TRIAL: NCT01784445
Title: Diclophenac Potassium Versus Ceftazidime for Reduction of Post ERCP Pancreatitis in Average Risk Patients-double Blind, Randomised Controlled Trial
Brief Title: Post ERCP Pancreatitis Prevention in Average Risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Rijeka (Other)
Responsible Party: Principal Investigator, Goran Hauser, Goran Hauser, MD, PhD, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PEP 2013
Record Dates: First submitted 2013-01-27; First posted 2013-02-05 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatitis
Keywords: Endoscopic Retrograde Cholangiopancreatography,
MeSH Terms: conditions — Pancreatitis | interventions — Ceftazidime

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftazidime plus placebo (Experimental): Procedure/Surgery: ERCP Each patient will receive: Ceftazidime 2 g i.v. once daily 30 minutes prior to procedure and glycerin suppository as placebo
  Interventions: Drug: Ceftazidime
- Diclophenac sodium plus placebo (Active Comparator): Procedure/Surgery:ERCP Each patient will receive 100 mg Diclophenac suppositories, once daily immediately prior to procedure plus 100 ml of saline as placebo
  Interventions: Drug: Ceftazidime

INTERVENTIONS:
Drug: Ceftazidime — Patient undergone ERCP will receive either diclophenac sodium suppositories(100mg)plus placebo or ceftazidime (2g i.v.) plus placebo before procedure
  Other Names: Fortaz

SUMMARY:
Diclophenac potassium and ceftazidime are commercially available drugs that are used in various clinical situations. They are safe and known for years. Diclophenac potassium and Ceftazidime have been used in some studies for the prophylaxis and treatment of pancreatitis and Post-ERCP Pancreatitis (PEP). Diclophenac potassium, together with indometacin is currently standard treatment for prevention of (PEP) while ceftazidime is possible alternative treatment for patients with contraindications for nonsteroidal medicines. The aim of the study is to evaluate the efficacy of Ceftazidime for the prophylaxis of PEP.

DETAILED DESCRIPTION:
Study type:

Interventional Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Parallel Assignment Masking: only Investigator Primary Purpose: Prevention Study Phase: Phase 4

Conditions or Focus of the study: Post ERCP pancreatitis

Intervention information

* Intervention Names ERCP
* Arm Information

  * Arm 1:Ceftazidime
  * Arm 2 (active comparator): Diclophenac potassium

ELIGIBILITY:
Inclusion Criteria:

* o All patients undergone to ERCP irrespectively about the diagnosis

Exclusion Criteria:

* o Unwillingness or inability to consent for the study

  * Age < 18 years
  * Previous ERCP (papillotomy)
  * Intrauterine pregnancy
  * Breast feeding mother
  * Allergy to Aspirin or NSAIDs and Ceftazidime
  * NSAID or antibiotic use within 1 week (ASA 325 mg daily or less acceptable)
  * Renal failure (Cr > 1.4)
  * Active or recent (within 4 weeks) gastrointestinal hemorrhage
  * Existing acute pancreatitis (lipase peak) within 72 hours prior to ERCP
  * Anticipated inability to follow protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of PEP in the group of patients receiving Ceftazidime versus incidence of PEP in the group of patients receiving Diclophenac potassium | One year

OTHER OUTCOMES:
Time to discharge from hospital | One year
  Influence of PEP severity on time to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Goran Hauser, MD, PhD, Principal Investigator — University Hospital Rijeka
Locations (1):
- Clinical Hospital Centre, Rijeka, Kresimirova 42, Croatia